CLINICAL TRIAL: NCT01744509
Title: PillCam Colon Capsule 2® (PCC2) in the Setting of Colorectal Cancer Screening (CRC) Program: Comparison With a New Integrated Reference Standard
Brief Title: PillCam Colon Capsule 2® (PCC2) in the Setting of Colorectal Cancer Screening Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Valduce Hospital (Other)
Responsible Party: Principal Investigator, Emanuele Rondonotti, MD, PhD, Valduce Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 25-2011
Record Dates: First submitted 2012-12-03; First posted 2012-12-06 (Estimated); Last update posted 2012-12-06 (Estimated); Status verified 2012-12

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnosis of CRC (Other): All the patients enrolled received all the 3 procedures: capsule colonoscopy; CT-colonography and optical colonoscopy.
  Interventions: Device: Capsule colonoscopy;

INTERVENTIONS:
Device: Capsule colonoscopy; — All the enrolled patients underwent all the three study procedures; the colon capsule is the intervention under evaluation; the other 2 procedures (Ct colonography and optcal colonoscopy contribute to build the composite reference standard)
  Other Names: Capsule colonoscopy: PillCam Coln Capsule 2

SUMMARY:
In this study the investigators evaluate the sensitivity of PCC2 (PillCam Colon Capsule 2 (R)) in identifying significant polyps in a CRC (Colo Recatal Cancer) screening program (primary outcome measure).

Each enrolled patient underwent three procedures: colon capsule endoscopy, CT-colonography and optical colonoscopy. In this study the reference standard is represented by the segmental unblinded colonoscopy (the unblinding is based on results of both capsule endoscopy and Ct colonography) The investigators also evaluated the tolerability of PCC2 as compared to optical colonoscopy (OC) and CT-colonography (CTC).

DETAILED DESCRIPTION:
Asymptomatic average risk subjects with positive iFOBT (immunochemical Fecal Occult Blood Test), participating the regional screening program, were offered to undergo PCC2 (PillCam Colon Capsule 2 (R)) followed, 21 days later, by CTC and OC performed on the same day. The number, size and location of significant polyps (>6mm) identified by each procedure were compared with the reference standard (RS), which was represented by the segmental unblinded colonoscopy. The unblinding was based on the integration of CTC and PCC2 results. For the PPC2 the quality of the bowel preparation (adequate/inadequate) and the completeness of the examination (capsule excreted still working or visualization of the anal verge) were also reported. In order to evaluate the tolerability, each subject was asked to identify, among the 3 procedures performed, which was the less tolerated one and which one he would be willing to repeat.

ELIGIBILITY:
Inclusion Criteria:

* asymptomatic average risk subjects, participating the regional colon cancer screening program, with positive iFOBT referred for colonoscopy

Exclusion Criteria:

* presence of obstructive symptoms
* swallowing disorders
* presence of cardiac pacemaker

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2011-03; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of PillCam Colon Capsule 2 (R) in identifying significant colonic polyps | participants are followed for about 1 month
  The number, size and location of significant polyps (>6mm) identified by each procedure were compared with the reference standard (RS), which was represented by the segmental unblinded colonoscopy.

SECONDARY OUTCOMES:
to evaluate the tolerability of PCC2 as compared to optical colonoscopy (OC) and CT-colonography (CTC). | participants are followed for about 1 month
  In order to evaluate the tolerability, each subject was asked to identify, among the 3 procedures performed, which was the less tolerated one and which one he would be willing to repeat.

CONTACTS AND LOCATIONS:
Overall Officials: Giancarlo Spinzi, Principal Investigator — Gastroenterology Unit; Ospedale Valduce
Locations (1):
- Ospedale Valduce, Como, Italy

REFERENCES:
- [Derived] Rondonotti E, Borghi C, Mandelli G, Radaelli F, Paggi S, Amato A, Imperiali G, Terreni N, Lenoci N, Terruzzi V, Baccarin A, Martegani A, Spinzi G. Accuracy of capsule colonoscopy and computed tomographic colonography in individuals with positive results from the fecal occult blood test. Clin Gastroenterol Hepatol. 2014 Aug;12(8):1303-10. doi: 10.1016/j.cgh.2013.12.027. Epub 2014 Jan 5. PMID 24398064